CLINICAL TRIAL: NCT00174109
Title: The Relation of Microtubule-Associated Protein 2 and Cell Migration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700625
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-06

CONDITIONS: Oral Cancer
Keywords: arecoline, oral cancer, MAP2, cell migration
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective

SUMMARY:
Clarify the relation of microtubule-associated protein 2 and cell migration

DETAILED DESCRIPTION:
Betel quid chewing has been shown to have intimate correlation with oral cancer. In Taiwan, the incidence of oral cancer is the fourth most common malignancy in male and in fact, 90% of which has been linked to betel quid chewing. The predisposing factors in oral cancers between the western countries and India, Southeast Asia including Taiwan are different. The factor is smoking in the former countries and betel quid chewing is the most important one in the latter groups. The genetic aberrations of oral cancers are different too between the western countries and India, Southeast Asia including Taiwan. The percentage of RAS mutations of oral cancers in the western countries is around 5%, and 35% in the India. In Taiwan, the RAS mutation rate revealed with immunohistochemical staining is 92%, comparing with those in western countries (62%), Japan (55-65%) and vice versa in the p53 mutations. The percentage of p53 mutations of oral cancers in the western countries is around 50%, and 16% in the India, Southeast Asia and Taiwan. It is generally believed that betel nut itself, arecoline and arecaidine, the major betel alkaloids, account for the etiological factors in the pathogenesis of oral cancer while betel quid supplements, unlike the former two main components, were reported to have little relevancy to oral cancer. Despite the fact that the cytotoxic and genotoxic effects of betel nut extract and arecoline, arecaidine have been extensively documented, and that some well-studied oncogenes or tumor suppressor genes have been implicated in betel quid-related oral cancer, the molecular mechanisms, addressed in a broader view, by which betel nut ingredients lead to oral tumorigenesis are not fully understood. Our preliminary results, by virtue of different genome-wide screening approaches to explore cellular functions of protein kinases in this context, identified several candidates that showed differential expression upon treatment of BQ on primary cultures from human oral mucosa. Of the candidates isolated, microtubule-associated protein 2 (MAP2), a neuron-specific cytoskeletal protein that is thought to predominantly express in rat brain cells, was found up-regulated at RNA level by RT-PCR in primary cultures. Our expanded immunohistochemical results of normal mucosa, leukoplakia and oral squamous cell carcinoma (OSCC) suggest that expression of the MAP2 significantly correlates with progression of BQ-induced OSCC (P = 0.0046), since the percentage of MAP2 positive staining is as much fourfold in BQ-exposed OSCC (41.2%) as in BQ-free OSCC (10.5%), whereas normal mucosa and leukoplakia show much less immunoreactivity as a whole. Furthermore, the MAP2 is shown to be preferentially expressed in histopathologically less differentiated OSCC (P = 0.014). Finally, we show that the MAP2 is highly expressed in the majority of invasive OSCC (67%). Consequently, this finding, in conjunction with the previous one, raise a possibility that overexpression of the MAP2 may play a critical role in the development of highly malignant OSCC characteristic of invasive and/or metastatic. Here we study the issue by establishing an in vitro system where extracts from the whole betel quid sandwiches are used to treat head and neck cancer cell lines and primary oral epithelial cells and subsequently, the effects of such treatments will be evaluated in terms of cell migration, Western blotting. Eight head and neck cancer cell lines and normal oral mucosae from 8 patients undergoing oral surgery will be collected. Extracts from the whole betel quid sandwiches with the concentration of 1.5 mg/ml will be added to the cell lines and primary oral epithelial cells for 1,3 and 5 days, respectively. Migration assay and detection of MAP2 expression will be performed to elucidate the relationship of MAP2 and cell migration.

ELIGIBILITY:
Inclusion Criteria:

* oral cancer

Exclusion Criteria:

* nil

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-08; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Jenq-Yuh Ko, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan